CLINICAL TRIAL: NCT01350804
Title: A Randomized, Double-blind, Placebo- and Active-controlled Study of Secukinumab to Demonstrate the Efficacy at 24 Weeks and to Assess the Safety, Tolerability and Long Term Efficacy up to 1 Year in Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Anti-TNFα Agents (CAIN457F2309) and A Four Year Extension Study to Evaluate the Long Term Efficacy, Safety and Tolerability of Secukinumab in Patients With Active Rheumatoid Arthritis (CAIN457F2309E1)
Brief Title: Efficacy at 24 Weeks and Safety, Tolerability and Long Term Efficacy of Secukinumab (AIN457) in Patients With Active Rheumatoid Arthritis (RA) and an Inadequate Response to Anti-Tumor Necrosis Factor α (Anti-TNFα) Agents (CAIN457F2309 and CAIN457F2309E1)
Acronym: NURTURE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F2309; 2011-000102-21 (EudraCT Number); NCT01640938 (obsolete NCT alias)
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-05

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; RA; ACR; inflammatory joints
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — secukinumab; Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- AIN457 10mg/kg - 75 mg (Experimental): Participants received AIN457 i.v. (10 mg/kg) at Baseline (BSL), Weeks 2 and 4 then AIN457 75 mg s.c. at Week 8 and injected every 4 weeks
  Interventions: Biological: AIN457
- AIN457 10mg/kg - 150 mg (Experimental): Participants received AIN457 i.v. (10 mg/kg) at BSL, Weeks 2 and 4 then AIN457 150 mg s.c. at Week 8 and injected every 4 weeks
  Interventions: Biological: AIN457
- Placebo (Placebo Comparator): Participants received matching placebo to AIN457 until week 16 or week 24 based on responder status (>= 20% reduction in tender and swollen joint count). Non-responders were switched to active treatment at week 16. Responders were switched to active treatment at week 24.
  Interventions: Biological: AIN457; Biological: Placebo
- Abatacept (Active Comparator): Participants received abatacept (from 500 to 1000 mg i.v. based on weight). Participants who did not respond to abatacept at Week 16 were re-randomized 1:1 to AIN457 75mg or 150mg at week 24 (after an 8 week washout period).
  Interventions: Biological: AIN457; Biological: Abatacept

INTERVENTIONS:
Biological: AIN457 — AIN457 (Secukinumab) is a human monoclonal antibody. Secukinumab binds and reduces the activity of Interleukin 17 (IL-17). AIN457 was given as i.v. (10mg/kg) at baseline, week 2 and week 4, and then s.c. (75 or 150mg) every 4 weeks starting at week 8.
  Other Names: Secukinumab
Biological: Placebo — Placebo was given as i.v. at baseline, week 2 and week 4, and then s.c. every 4 weeks starting at week 8.
  Arms: Placebo
Biological: Abatacept — Abatacept (from 500 to 1000 mg i.v. based on weight) was given as i.v. at baseline, weeks 2 and 4, and then every 4 weeks starting at week 8.
  Other Names: Orencia
  Arms: Abatacept

SUMMARY:
The core and extension studies assessed the safety and efficacy of secukinumab when added to a background therapy in patients with active rheumatoid arthritis who are intolerant to or have had an inadequate response to anti-TNF-α agents. Patients received either secukinumab, placebo or abatacept (active comparator). The core study was completed. However, the extension study was prematurely terminated after the primary endpoint analysis of the core study at week 24 had demonstrated numerically higher efficacy for the active comparator abatacept compared to secukinumab.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female patients
* Presence of RA classified by ACR 2010 revised criteria for at least 3 months before screening
* At Baseline: Disease activity criteria defined by >= 6 tender joints out of 68 and >= 6 swollen joints out of 66

WITH at least 1 of the following at screening:

* Anti-Cyclic Citrullinated Peptide (Anti-CCP) antibodies positive OR
* Rheumatoid Factor positive

AND WITH at least 1 of the following at screening:

* High sensitivity C-Reactive Protein (hsCRP) >= 10 mg/L OR
* Erythrocyte Sedimentation Rate (ESR) >= 28 millimeter (mm)/1st hour
* Patients must have been taking at least one anti-TNF-α agent given at an approved dose for at least 3 months before randomization and have experienced an inadequate response to treatment or have been intolerant to at least one administration of an anti-TNF-α agent
* Patients must be taking MTX or any other DMARD (but not more than 1 DMARD) for at least 3 months before randomization and have to be on a stable dose at least 4 weeks before randomization (7.5 to 25 mg/week for MTX or other DMARD at maximum tolerated dose)

Exclusion Criteria:

* Chest x-ray with evidence of ongoing infectious or malignant process, obtained within 3 months prior to screening and evaluated by a qualified physician
* RA patients functional status class IV according to the ACR 1991 revised criteria
* Patients who have ever received biologic immunomodulating agents except for those targeting TNFα
* Previous treatment with any cell-depleting therapies

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2011-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (107):
- United States (43):
  - Novartis Investigative Site, Anniston, Alabama
  - Novartis Investigative Site, Vestavia Hills, Alabama
  - Novartis Investigative Site, Freemont, California
  - Novartis Investigative Site, Pomona, California
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Van Nuys, California
  - Novartis Investigative Site, Bridgeport, Connecticut
  - Novartis Investigative Site, Aventura, Florida
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Hialeah, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Palm Harbor, Florida
  - Novartis Investigative Site, Pembroke Pines, Florida
  - Novartis Investigative Site, Pensacola, Florida
  - Novartis Investigative Site, Plantation, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Coeur d'Alene, Idaho
  - Novartis Investigative Site, Morton Grove, Illinois
  - Novartis Investigative Site, Springfield, Illinois
  - Novartis Investigative Site, Wichita, Kansas
  - Novartis Investigative Site, Bowling Green, Kentucky
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Lansing, Michigan
  - Novartis Investigative Site, Eagan, Minnesota
  - Novartis Investigative Site, Kansas City, Missouri
  - Novartis Investigative Site, Richmond Heights, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Zanesville, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Jackson, Tennessee
  - Novartis Investigative Site, Kingsport, Tennessee
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Carrollton, Texas
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Sugar Land, Texas
  - Novartis Investigative Site, Waco, Texas
  - Novartis Investigative Site, Spokane, Washington
  - Novartis Investigative Site, Clarksburg, West Virginia
- Brazil (4):
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Bulgaria (4):
  - Novartis Investigative Site, Plovdiv, Bulgaria
  - Novartis Investigative Site, Rousse, Bulgaria
  - Novartis Investigative Site, Sevlievo, Bulgaria
  - Novartis Investigative Site, Sofia, Bulgaria
- Canada (3):
  - Novartis Investigative Site, St. John's, Newfoundland and Labrador
  - Novartis Investigative Site, Sainte-Foy, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Colombia (3):
  - Novartis Investigative Site, Bogotá, Cundinamarca
  - Novartis Investigative Site, Barranquilla
  - Novartis Investigative Site, Bogotá
- Czechia (4):
  - Novartis Investigative Site, Bruntál, Czech Republic
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Uherské Hradiště, Czech Republic
  - Novartis Investigative Site, Zlín, Czech Republic
- France (5):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Cahors
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Germany (12):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Cottbus
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Gommern
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Zerbst
- Hungary (4):
  - Novartis Investigative Site, Győr, Hungary
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Gyula
  - Novartis Investigative Site, Szolnok
- Italy (5):
  - Novartis Investigative Site, Valeggio sul Mincio, (vr)
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Siena, SI
- Mexico (5):
  - Novartis Investigative Site, Mexicali, Estado de Baja California
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Monterrey, Nuevo León
  - Novartis Investigative Site, Culiacán, Sinaloa
- Novartis Investigative Site, Iași, Iaşi, Romania
- Russia (5):
  - Novartis Investigative Site, Korolyov
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Tula
- Slovakia (2):
  - Novartis Investigative Site, Banská Bystrica, Slovak Republic
  - Novartis Investigative Site, Piešťany, Slovakia
- Spain (7):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid, Madrid

REFERENCES:
- [Derived] Huang Y, Fan Y, Liu Y, Xie W, Zhang Z. Efficacy and safety of secukinumab in active rheumatoid arthritis with an inadequate response to tumor necrosis factor inhibitors: a meta-analysis of phase III randomized controlled trials. Clin Rheumatol. 2019 Oct;38(10):2765-2776. doi: 10.1007/s10067-019-04595-1. Epub 2019 May 14. PMID 31087226
- [Derived] Blanco FJ, Moricke R, Dokoupilova E, Codding C, Neal J, Andersson M, Rohrer S, Richards H. Secukinumab in Active Rheumatoid Arthritis: A Phase III Randomized, Double-Blind, Active Comparator- and Placebo-Controlled Study. Arthritis Rheumatol. 2017 Jun;69(6):1144-1153. doi: 10.1002/art.40070. Epub 2017 May 3. PMID 28217871

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At baseline, participants were randomized to 1 of 4 treatment groups. Placebo non-responders at week16 were re-randomized to receive AIN457 75mg or AIN457 150mg. Placebo responders at Week16 were re-randomized to receive AIN457 75mg or AIN457 150mg at Week24. Fifteen participants from the placebo group discontinued prior to re-randomization.
Pre-assignment Details: Abatacept responders at Week16 continued on abatacept and non-responders at Week 16 were re-randomized to begin either AIN457 75mg or AIN457 150mg at Week 24. Of the 551 core study participants, 254 participants entered the extension study.
Period: Core Study
Arm/Group | AIN457 10mg/kg - 75 mg | AIN457 10mg/kg - 150 mg | Placebo | Abatacept
Started | 138 | 137 | 138 | 138
Safety Set | 137 (1 participant actually received placebo; participant was reassigned to placebo for safety analysis.) | 136 (1 participant did not receive treatment; therefore participant was not counted in safety analysis.) | 139 (1 participant actually received placebo; participant was reassigned to placebo for safety analysis.) | 137 (1 participant did not receive treatment; therefore participant was not counted in safety analysis.)
Tratment Switch to AIN457 at Week 16 | 0 | 0 | 78 (15 participantsdiscontinued prior to the treatment switch) | 0
Treatment Switch to AIN457 at Week 24 | 0 | 0 | 45 | 37
Full Analysis Set | 138 | 137 | 138 | 138
Completed | 97 | 90 | 91 | 112
Not Completed | 41 | 47 | 47 | 26
Not completed — Withdrawal by Subject | 11 | 17 | 16 | 7
Not completed — Study terminated by Sponsor | 0 | 0 | 0 | 2
Not completed — Protocol deviation | 1 | 0 | 1 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 3
Not completed — Lost to Follow-up | 3 | 0 | 2 | 1
Not completed — Lack of Efficacy | 16 | 19 | 18 | 5
Not completed — Death | 1 | 1 | 1 | 0
Not completed — Adverse Event | 8 | 10 | 8 | 8
Period: Extension Study, Weeks 52 - 260
Arm/Group | AIN457 10mg/kg - 75 mg | AIN457 10mg/kg - 150 mg | Placebo | Abatacept
Started | 80 | 79 | 72 (During the extension, these participants received AIN457.) | 23 (During the extension, these participants received AIN457.)
Completed | 0 | 0 | 0 | 0
Not Completed | 80 | 79 | 72 | 23
Not completed — Withdrawal by Subject | 5 | 6 | 4 | 3
Not completed — Study terminated by Sponsor | 67 | 67 | 64 | 16
Not completed — Physician Decision | 1 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 4 | 4 | 0 | 1
Not completed — Adverse Event | 3 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 10mg/kg - 75 mg | AIN457 10mg/kg - 150 mg | Placebo | Abatacept | Total
Number analyzed (Participants) | 138 | 137 | 138 | 138 | 551
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 111 | 103 | 106 | 115 | 435
  >=65 years | 27 | 34 | 32 | 23 | 116
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 109 | 115 | 107 | 450
  Male | 19 | 28 | 23 | 31 | 101

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an American College of Rheumatology Response 20 (ACR20).
Description: ACR20 response was defined as having a positive clinical response to treatment (individual improvement) in disease activity if the participant had at least 20% improvement in tender 68-joint count, swollen 66-joint count and at least 3 of the following 5 measures: patient's assessment of RA pain, patient's global assessment of disease activity, physician's global assessment of disease activity, subject self-assessed disability (Health Assessment Questionnaire [HAQ-DI] score), and/or acute phase reactant (high sensitivity c-reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR). The ACR20 response results at week 24 used non-responder imputation.
Time Frame: week 24
Population: Full analysis set: the full analysis set was comprised of all randomized participants (excluding mis-randomized participants) who were assigned to study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 10mg/kg - 75 mg | AIN457 10mg/kg - 150 mg | Placebo | Abatacept
Number analyzed (Participants) | 138 | 137 | 138 | 138
Percentage of participants | 28.3 | 30.7 | 18.1 | 42.8
Statistical Analysis 1: Comparison: AIN457 10mg/kg - 75 mg vs Placebo; Test type: Superiority or Other; p = 0.0458, Regression, Logistic; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.0 to 3.2]
Statistical Analysis 2: Comparison: AIN457 10mg/kg - 150 mg vs Placebo; Test type: Superiority or Other; p = 0.0152, Regression, Logistic; Odds Ratio (OR) = 2.02, 95% CI 2-sided [1.1 to 3.5]

2. Secondary Outcome: Change From Baseline in Disease Activity Score Utilizing CRP (DAS28-CRP)
Description: The DAS28 is a measure of disease activity in RA based on Swollen and Tender Joint Counts (out of a total of 28), hsCRP and the Patient's Global Assessment of Disease Activity. A DAS28 score greater than 5.1 implies active disease, equal to or less than 3.2 low disease activity, and less than 2.6 remission. A negative change from baseline indicates improvement.
Time Frame: baseline, week 24
Population: Participants from the full analysis set were considered for the analysis. Participants with measurements at both baseline and week 24 were analyzed. The full analysis set was comprised of all randomized participants (excluding mis-randomized participants) who were assigned to study treatment.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AIN457 10mg/kg - 75 mg | AIN457 10mg/kg - 150 mg | Placebo | Abatacept
Number analyzed (Participants) | 116 | 108 | 44 | 84
score on a scale | -1.47 (0.115) | -1.47 (0.119) | -1.02 (0.163) | -2.07 (0.128)

3. Secondary Outcome: Change From Baseline in Stanford Health Assessment Questionnaire Disability Index (HAQ-DI)
Description: The HAQ-DI assesses a subject's level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities. There are 20 questions in 8 categories of functioning including dressing, rising, eating, walking, hygiene, reach, grip and usual activities. The stem of each item asks 'Over the past week, "are you able to..." perform a particular task'. Each item is scored on a 4 point scale from 0 - 3, representing normal, no difficulty (0), some difficulty (1), much difficulty (2) and unable to do (3). The disability index score is calculated as the mean of the available category scores, ranging from 0 to 3. A negative change from baseline indicates improvement.
Time Frame: baseline, week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AIN457 10mg/kg - 75 mg | AIN457 10mg/kg - 150 mg | Placebo | Abatacept
Number analyzed (Participants) | 117 | 110 | 44 | 86
score on a scale | -0.30 (0.049) | -0.39 (0.051) | -0.26 (0.065) | -0.61 (0.053)

4. Secondary Outcome: Percentage of Participants Achieving ACR50
Description: ACR50 response was defined as having a positive clinical response to treatment (individual improvement) in disease activity if the participant had at least 50% improvement in tender 68-joint count, swollen 66-joint count and at least 3 of the following 5 measures: patient's assessment of RA pain, patient's global assessment of disease activity, physician's global assessment of disease activity, subject self-assessed disability (Health Assessment Questionnaire [HAQ-DI] score), and/or acute phase reactant (high sensitivity c-reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR). The ACR50 response results at week 24 used non-responder imputation.
Time Frame: week 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 10mg/kg - 75 mg | AIN457 10mg/kg - 150 mg | Placebo | Abatacept
Number analyzed (Participants) | 138 | 137 | 138 | 138
Percentage of participants | 11.6 | 16.8 | 9.4 | 27.5

5. Secondary Outcome: Percentage of Participants Achieving ACR20, ACR 50 and ACR 70 - Using Non-responder Imputation
Description: ACR20, ACR 50 and ACR 70 response was defined as having a positive clinical response to treatment (individual improvement) in disease activity if the participant had at least 20%, 50% and/or 70% improvement, respectively, in tender 68-joint count, swollen 66-joint count and at least 3 of the following 5 measures: patient's assessment of RA pain, patient's global assessment of disease activity, physician's global assessment of disease activity, subject self-assessed disability (Health Assessment Questionnaire [HAQ-DI] score), and/or acute phase reactant (high sensitivity c-reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR).
Time Frame: baseline, weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: Participants from the full analysis set were considered for the analysis. Participants with missing data were considered non-responders at the respective time point. Placebo and Abatacept participants were considered non-responders from the time of treatment switch.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 10mg/kg - 75 mg | AIN457 10mg/kg - 150 mg | Placebo | Abatacept
Number analyzed (Participants) | 138 | 137 | 138 | 138
Percentage of participants
  ACR20, week 1 | 21.0 | 17.5 | 7.2 | 10.9
  ACR20, week 2 | 24.6 | 21.2 | 12.3 | 23.9
  ACR20, week 4 | 34.1 | 27.0 | 21.7 | 31.2
  ACR20, week 8 | 35.5 | 41.6 | 21.0 | 49.3
  ACR20, week 12 | 28.3 | 33.6 | 24.6 | 47.1
  ACR20, week 16 | 34.1 | 39.4 | 23.2 | 51.4
  ACR20, week 20 | 26.8 | 38.0 | 18.1 | 47.8
  ACR20, week 24 | 28.3 | 30.7 | 18.1 | 42.8
  ACR50, week 1 | 6.5 | 2.9 | 0.7 | 1.4
  ACR50, week 2 | 5.1 | 8.8 | 2.9 | 2.9
  ACR50, week 4 | 9.4 | 10.2 | 2.9 | 7.2
  ACR50, week 8 | 7.2 | 15.3 | 10.1 | 18.8
  ACR50, week 12 | 8.7 | 13.1 | 10.1 | 22.5
  ACR50, week 16 | 13.8 | 20.4 | 9.4 | 23.9
  ACR50, week 20 | 12.3 | 18.2 | 8.0 | 26.8
  ACR50, week 24 | 11.6 | 16.8 | 9.4 | 27.5
  ACR70, week 1 | 0.7 | 0.7 | 0.0 | 0.7
  ACR70, week 2 | 1.4 | 0.7 | 1.4 | 0.7
  ACR70, week 4 | 4.3 | 2.9 | 1.4 | 1.4
  ACR70, week 8 | 1.4 | 4.4 | 2.9 | 5.8
  ACR70, week 12 | 2.2 | 2.9 | 2.9 | 9.4
  ACR70, week 16 | 5.1 | 8.0 | 2.9 | 9.4
  ACR70, week 20 | 4.3 | 7.3 | 5.8 | 10.1
  ACR70, week 24 | 5.1 | 10.2 | 5.1 | 12.3

6. Secondary Outcome: Percentage of Participants Achieving ACR20, ACR 50 and ACR 70 - Observed Data
Description: ACR20, ACR 50 and ACR 70 response was defined as having a positive clinical response to treatment (individual improvement) in disease activity if the participant had at least 20%, 50% and/or 70% improvement, respectively, in tender 68-joint count, swollen 66-joint count and at least 3 of the following 5 measures: patient's assessment of RA pain, patient's global assessment of disease activity, physician's global assessment of disease activity, subject self-assessed disability (Health Assessment Questionnaire [HAQ-DI] score), and/or acute phase reactant (high sensitivity c-reactive protein (hsCRP) or erythrocyte sedimentation rate (ESR). The ACR20, ACR50 and ACR70 response results from baseline up to week 52 were based on observed data, i.e. without imputation.
Time Frame: baseline, weeks 1, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: Participants from the full analysis set were considered for the analysis. Participants with measurements at both baseline and each post-baseline time point were analyzed for that post-baseline time point. The full analysis set was comprised of all randomized participants (excluding mis-randomized participants) who were assigned to study treatment.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo Non-responder - AIN457 75 mg: Participants switched from placebo to AIN457 75 mg starting at week 16.
- Placebo Non-responder - AIN457 150 mg: Participants switched from placebo to AIN457 150 mg starting at week 16.
- Placebo Responder - AIN457 75mg: Participants switched from placebo to AIN457 75 mg starting at week 24.
- Placebo Responder - AIN457 150mg: Participants switched from placebo to AIN457 150 mg starting at week 24.
- Abatacept Responders: Abatacept responders remained on abatacept (from 500 to 1000 mg iv based on weight).
- Abatacept Non-respnders - AIN457 75mg: Participants switched from abatacept to AIN457 75 mg starting at week 24.
- Abatacept Non-responders - AIN457 150mg: Participants switched from abatacept to AIN457 150 mg starting at week 24.
Arm/Group | AIN457 10mg/kg - 75 mg | AIN457 10mg/kg - 150 mg | Placebo | Abatacept | Placebo Non-responder - AIN457 75 mg | Placebo Non-responder - AIN457 150 mg | Placebo Responder - AIN457 75mg | Placebo Responder - AIN457 150mg | Abatacept Responders | Abatacept Non-respnders - AIN457 75mg | Abatacept Non-responders - AIN457 150mg
Number analyzed (Participants) | 138 | 137 | 138 | 138 | 39 | 39 | 23 | 22 | 101 | 18 | 19
Percentage of participants
  ACR20,wk 1,n=132,129,130,130,39,35,21,22,96,17,17 | 22.7 | 18.6 | 7.7 | 11.5 | 5.1 | 5.7 | 14.3 | 13.6 | 14.6 | 0.0 | 5.9
  ACR20,wk 2,n=131,130,134,134,39,36,23,22,99,17,18 | 26.7 | 22.3 | 12.7 | 25.4 | 2.6 | 11.1 | 34.8 | 13.6 | 29.3 | 11.8 | 16.7
  ACR20,wk 4,n=133,132,131,129,39,39,23,21,93,17,19 | 36.1 | 28.0 | 22.9 | 34.1 | 15.4 | 12.8 | 43.5 | 42.9 | 41.9 | 17.6 | 10.5
  ACR20,wk 8,n=132,127,131,131,39,39,23,22,95,17,19 | 38.6 | 44.9 | 22.1 | 52.7 | 17.9 | 12.8 | 39.1 | 31.8 | 61.1 | 29.4 | 31.6
  ACR20,wk 12,n=130,115,123,129,39,37,23,21,94,17,18 | 30.8 | 40.0 | 27.6 | 51.2 | 15.4 | 16.2 | 47.8 | 52.4 | 62.8 | 17.6 | 22.2
  ACR20,wk 16,n=126,118,116,129,36,37,21,22,94,16,19 | 38.1 | 45.8 | 27.6 | 55.8 | 2.8 | 2.7 | 76.2 | 63.6 | 76.6 | 0.0 | 0.0
  ACR20,wk 20,n=122,114,119,126,38,37,23,21,91,16,19 | 39.3 | 51.8 | 42.9 | 57.9 | 42.1 | 29.7 | 60.9 | 47.6 | 73.6 | 6.3 | 26.3
  ACR20,wk 24,n=117,110,117,121,38,36,21,22,87,16,18 | 45.3 | 48.2 | 40.2 | 57.9 | 26.3 | 33.3 | 57.1 | 59.1 | 69.0 | 31.3 | 27.8
  ACR20,wk28,n=115,103,na,na,33,35,21,21,86,17,19 | 47.8 | 65.0 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 33.3 | 37.1 | 71.4 | 90.5 | 74.4 | 41.2 | 42.1
  ACR20,wk32,n=104,97,na,na,33,30,21,19,87,17,17 | 56.7 | 61.9 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 51.5 | 36.7 | 81.0 | 68.4 | 74.7 | 23.5 | 47.1
  ACR20,wk36,n=102,93,na,na,30,30,21,20,85,18,16 | 56.9 | 53.8 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 46.7 | 56.7 | 85.7 | 65.0 | 77.6 | 27.8 | 56.3
  ACR20,wk40,n=96,90,na,na,28,28,21,19,85,15,17 | 53.1 | 61.1 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 53.6 | 53.6 | 85.7 | 73.7 | 71.8 | 40.0 | 58.8
  ACR20,wk44,n=97,90,na,na,28,27,20,18,84,15,16 | 56.7 | 61.1 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 50.0 | 55.6 | 85.0 | 77.8 | 77.4 | 33.3 | 31.3
  ACR20,wk48,n=94,89,na,na,28,26,18,19,77,12,14 | 57.4 | 68.5 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 53.6 | 61.5 | 72.2 | 57.9 | 71.4 | 25.0 | 50.0
  ACR20,wk52,n=92,88,na,na,28,26,20,18,79,15,15 | 56.5 | 62.5 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 39.3 | 57.7 | 75.0 | 88.9 | 74.7 | 40.0 | 33.3
  ACR50,wk1,n=132,129,130,130,39,35,21,22,96,17,17 | 6.8 | 3.1 | 0.8 | 1.5 | 0.0 | 0.0 | 4.8 | 0.0 | 1.0 | 0.0 | 5.9
  ACR50,wk2,n=131,130,134,134,39,36,23,22,99,17,18 | 5.3 | 9.2 | 3.0 | 3.0 | 0.0 | 0.0 | 13.0 | 4.5 | 3.0 | 0.0 | 5.6
  ACR50,wk4,n=133,132,131,129,39,39,23,21,93,17,19 | 9.8 | 10.6 | 3.1 | 7.8 | 0.0 | 0.0 | 8.7 | 9.5 | 10.8 | 0.0 | 0.0
  ACR50,wk8,n=132,127,131,131,39,39,23,22,95,17,19 | 9.1 | 16.5 | 10.7 | 20.6 | 5.1 | 5.1 | 34.8 | 9.1 | 25.3 | 11.8 | 5.3
  ACR50,wk12,n=130,115,123,129,39,37,23,21,94,17,18 | 10.0 | 15.7 | 11.4 | 24.8 | 2.6 | 8.1 | 21.7 | 23.8 | 30.9 | 5.9 | 11.1
  ACR50,wk16,n=126,118,116,129,36,37,21,22,94,16,19 | 15.9 | 23.7 | 11.2 | 26.4 | 0.0 | 0.0 | 38.1 | 22.7 | 36.2 | 0.0 | 0.0
  ACR50,wk20,n=122,114,119,126,38,37,23,21,91,16,19 | 15.6 | 21.9 | 12.6 | 31.7 | 7.9 | 2.7 | 34.8 | 14.3 | 40.7 | 0.0 | 15.8
  ACR50,wk24,n=117,110,117,121,38,36,21,22,87,16,18 | 14.5 | 22.7 | 14.5 | 33.1 | 0.0 | 11.1 | 38.1 | 22.7 | 44.8 | 0.0 | 5.6
  ACR50,wk28,n=115,103,na,na,33,35,21,21,86,17,19 | 13.9 | 31.1 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 6.1 | 8.6 | 33.3 | 33.3 | 41.9 | 23.5 | 0.0
  ACR50,wk32,n=104,97,na,na,33,30,21,19,87,17,17 | 21.2 | 32.0 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 6.1 | 13.3 | 42.9 | 31.6 | 47.1 | 5.9 | 0.0
  ACR50,wk36,n=102,93,na,na,30,30,21,20,85,18,16 | 23.5 | 24.7 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 16.7 | 16.7 | 28.6 | 20.0 | 47.1 | 16.7 | 18.8
  ACR50,wk40,n=96,90,na,na,28,28,21,19,85,15,17 | 25.0 | 25.6 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 14.3 | 28.6 | 38.1 | 26.3 | 45.9 | 20.0 | 5.9
  ACR50,wk44,n=97,90,na,na,28,27,20,18,84,15,16 | 27.8 | 30.0 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 7.1 | 29.6 | 35.0 | 33.3 | 50.0 | 13.3 | 6.3
  ACR50,wk48,n=94,89,na,na,28,26,18,19,77,12,14 | 25.5 | 42.7 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 14.3 | 23.1 | 38.9 | 26.3 | 48.1 | 0.0 | 0.0
  ACR50,wk52,n=92,88,na,na,28,26,20,18,79,15,15 | 26.1 | 45.5 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 10.7 | 26.9 | 40.0 | 44.4 | 51.9 | 20.0 | 13.3
  ACR70,wk1,n=132,129,130,130,39,35,21,22,96,17,17 | 0.8 | 0.8 | 0.0 | 0.8 | 0.0 | 0.0 | 0.0 | 0.0 | 1.0 | 0.0 | 0.0
  ACR70,wk2,n=131,130,134,134,39,36,23,22,99,17,18 | 1.5 | 0.8 | 1.5 | 0.7 | 0.0 | 0.0 | 4.3 | 4.5 | 1.0 | 0.0 | 0.0
  ACR70,wk4,n=133,132,131,129,39,39,23,21,93,17,19 | 4.5 | 3.0 | 1.5 | 1.6 | 0.0 | 0.0 | 4.3 | 4.8 | 2.2 | 0.0 | 0.0
  ACR70,wk8,n=132,127,131,131,39,39,23,22,95,17,19 | 1.5 | 4.7 | 3.1 | 6.1 | 0.0 | 2.6 | 13.0 | 0.0 | 7.4 | 5.9 | 0.0
  ACR70,wk12,n=130,115,123,129,39,37,23,21,94,17,18 | 3.1 | 3.5 | 3.3 | 10.9 | 0.0 | 0.0 | 13.0 | 4.8 | 14.9 | 0.0 | 0.0
  ACR70,wk16,n=126,118,116,129,36,37,21,22,94,16,19 | 6.3 | 9.3 | 3.4 | 10.0 | 0.0 | 0.0 | 14.3 | 4.5 | 13.8 | 0.0 | 0.0
  ACR70,wk20,n=122,114,119,126,38,37,23,21,91,16,19 | 6.6 | 8.8 | 6.7 | 11.1 | 0.0 | 0.0 | 21.7 | 14.3 | 15.4 | 0.0 | 0.0
  ACR70,wk24,n=117,110,117,121,38,36,21,22,87,16,18 | 6.0 | 12.7 | 8.5 | 14.9 | 0.0 | 8.3 | 23.8 | 9.1 | 19.5 | 0.0 | 5.6
  ACR70,wk28,n=115,103,na,na,33,35,21,21,86,17,19 | 6.1 | 17.5 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 0.0 | 2.9 | 14.3 | 14.3 | 17.4 | 5.9 | 0.0
  ACR70,wk32,n=104,97,na,na,33,30,21,19,87,17,17 | 4.8 | 10.0 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 0.0 | 3.3 | 19.0 | 0.0 | 21.8 | 0.0 | 0.0
  ACR70,wk36,n=102,93,na,na,30,30,21,20,85,18,16 | 5.9 | 11.8 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 3.3 | 0.0 | 23.8 | 0.0 | 23.5 | 11.1 | 0.0
  ACR70,wk40,n=96,90,na,na,28,28,21,19,85,15,17 | 8.3 | 11.1 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 7.1 | 10.7 | 19.0 | 10.5 | 21.2 | 13.3 | 0.0
  ACR70,wk44,n=97,90,na,na,28,27,20,18,84,15,16 | 12.4 | 18.9 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 0.0 | 11.1 | 25.0 | 11.1 | 26.2 | 6.7 | 0.0
  ACR70,wk48,n=94,89,na,na,28,26,18,19,77,12,14 | 9.6 | 20.2 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 3.6 | 15.4 | 33.3 | 10.5 | 27.3 | 0.0 | 0.0
  ACR70,wk52,n=92,88,na,na,28,26,20,18,79,15,15 | 6.5 | 19.3 | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | 0.0 | 7.7 | 30.0 | 16.7 | 22.8 | 13.3 | 0.0

7. Secondary Outcome: Change From Baseline in HAQ-DI - Using Mixed Model Repeated Measures (MMRM)
Description: The HAQ-DI, assesses a subject's level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities. There are 20 questions in 8 categories of functioning including dressing, rising, eating, walking, hygiene, reach, grip and usual activities. The stem of each item asks 'Over the past week, "are you able to..." perform a particular task'. Each item is scored on a 4 point scale from 0 - 3, representing normal, no difficulty (0), some difficulty (1), much difficulty (2) and unable to do (3). The disability index score is calculated as the mean of the available category scores, ranging from 0 to 3. A negative change from baseline indicates improvement.
Time Frame: baseline, weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: Participants from the full analysis set were considered for this analysis. For Placebo and Abatacept participants, data collected after treatment switch was treated as missing, as were missing values for all treatment groups.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AIN457 10mg/kg - 75 mg | AIN457 10mg/kg - 150 mg | Placebo | Abatacept
Number analyzed (Participants) | 138 | 137 | 138 | 138
score on a scale
  week 1, n=132,129,130,129 | -0.22 (0.032) | -0.21 (0.032) | -0.08 (0.032) | -0.19 (0.032)
  week 2, n=131,130,134,133 | -0.22 (0.036) | -0.25 (0.036) | -0.16 (0.036) | -0.26 (0.036)
  week 4, n=133,133,131,130 | -0.30 (0.039) | -0.31 (0.040) | -0.17 (0.040) | -0.36 (0.040)
  week 8, n=132,127,131,130 | -0.29 (0.042) | -0.32 (0.043) | -0.17 (0.043) | -0.46 (0.043)
  week 12, n=130,114,123,129 | -0.31 (0.046) | -0.33 (0.047) | -0.18 (0.047) | -0.51 (0.046)
  week 16, n=127,118,116,129 | -0.30 (0.048) | -0.37 (0.049) | -0.22 (0.049) | -0.52 (0.048)
  week 20, n=122,114,47,92 | -0.36 (0.051) | -0.42 (0.052) | -0.21 (0.066) | -0.57 (0.054)
  week 24, n=117,110,44,86 | -0.30 (0.049) | -0.39 (0.051) | -0.26 (0.065) | -0.61 (0.053)

8. Secondary Outcome: Change From Baseline in HAQ-DI - Observed Data
Description: The HAQ-DI assesses a subject's level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities. There are 20 questions in 8 categories of functioning including dressing, rising, eating, walking, hygiene, reach, grip and usual activities. The stem of each item asks 'Over the past week, "are you able to..." perform a particular task'. Each item is scored on a 4 point scale from 0 - 3, representing normal, no difficulty (0), some difficulty (1), much difficulty (2) and unable to do (3). The disability index score is calculated as the mean of the available category scores, ranging from 0 to 3. A negative change from baseline indicates improvement. The HAQ-DI results from baseline up to week 52 were based on observed data, i.e. without imputation.
Time Frame: baseline, weeks 1, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo Non-responder - AIN457 75mg: Participants switched from placebo to AIN457 75 mg starting at week 16.
- Placebo Non-responder - AIN457 150mg: Participants switched from placebo to AIN457 150 mg starting at week 16.
- Abatacept Non-responders - AIN457 75mg: Participants switched from placebo to AIN457 75 mg starting at week 24.
Arm/Group | AIN457 10mg/kg - 75 mg | AIN457 10mg/kg - 150 mg | Placebo | Abatacept | Placebo Non-responder - AIN457 75mg | Placebo Non-responder - AIN457 150mg | Placebo Responder - AIN457 75mg | Placebo Responder - AIN457 150mg | Abatacept Responders | Abatacept Non-responders - AIN457 75mg | Abatacept Non-responders - AIN457 150mg
Number analyzed (Participants) | 138 | 137 | 138 | 138 | 39 | 39 | 23 | 22 | 101 | 18 | 19
score on a scale
  wk1,n=132,129,130,129,39,35,21,22,95,17,17 | -0.225 (0.3766) | -0.215 (0.4095) | -0.101 (0.3186) | -0.194 (0.4290) | -0.119 (0.2896) | -0.079 (0.3093) | -0.125 (0.4257) | -0.153 (0.2468) | -0.232 (0.4551) | -0.081 (0.3616) | -0.096 (0.3047)
  Wk2,n=131,130,134,133,39,36,23,22,133,98,17,18 | -0.215 (0.3877) | -0.239 (0.4885) | -0.191 (0.4340) | -0.254 (0.4520) | -0.122 (0.2605) | -0.176 (0.4631) | -0.380 (0.5063) | -0.250 (0.5015) | -0.300 (0.4693) | -0.132 (0.3630) | -0.118 (0.3987)
  Wk4,n=133,133,131,130,39,39,23,21,94,17,19 | -0.299 (0.4551) | -0.300 (0.5184) | -0.214 (0.4492) | -0.368 (0.5130) | -0.077 (0.3634) | -0.224 (0.4968) | -0.364 (0.5627) | -0.310 (0.3103) | -0.445 (0.5245) | -0.110 (0.3505) | -0.217 (0.4874)
  Wk8,n=132,127,131,130,39,39,23,22,94,17,19 | -0.277 (0.5062) | -0.309 (0.5175) | -0.217 (0.5457) | -0.463 (0.5182) | -0.186 (0.5097) | -0.128 (0.5077) | -0.543 (0.6313) | -0.176 (0.4782) | -0.543 (0.5289) | -0.206 (0.4900) | -0.303 (0.3780)
  wk12,n=130,114,123,129,39,37,23,21,94,17,18 | -0.287 (0.5384) | -0.307 (0.5488) | -0.241 (0.5152) | -0.508 (0.6369) | -0.109 (0.4783) | -0.179 (0.5133) | -0.451 (0.6167) | -0.381 (0.3982) | -0.622 (0.6520) | -0.221 (0.4274) | -0.181 (0.5376)
  Wk16,n=127,118,116,129,36,37,21,22,94,16,19 | -0.294 (0.5236) | -0.355 (0.6217) | -0.279 (0.5493) | -0.535 (0.6418) | -0.167 (0.5295) | -0.111 (0.4591) | -0.565 (0.5356) | -0.472 (0.5988) | -0.660 (0.6590) | -0.195 (0.4281) | -0.204 (0.4827)
  Wk20,n=122,114,119,125,38,37,23,21,90,16,19 | -0.333 (0.5111) | -0.402 (0.6429) | -0.319 (0.5637) | -0.583 (0.6654) | -0.237 (0.4756) | -0.179 (0.5158) | -0.543 (0.5325) | -0.470 (0.7309) | -0.699 (0.6849) | -0.086 (0.3972) | -0.454 (0.5436)
  Wk24,n=117,110,117,120,38,36,21,22,86,16,18 | -0.268 (0.4930) | -0.405 (0.5767) | 0.346 (0.5941) | -0.590 (0.6872) | -0.257 (0.4730) | -0.253 (0.6502) | -0.589 (0.5648) | -0.420 (0.6732) | -0.744 (0.6787) | -0.180 (0.4257) | -0.215 (0.6443)
  Wk28,n=115,102,na,na,33,35,21,21,86,17,19 | -0.304 (0.5342) | -0.439 (0.5780) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -0.345 (0.5880) | -0.336 (0.5846) | -0.625 (0.4809) | -0.601 (0.5571) | -0.689 (0.6428) | -0.309 (0.5522) | -0.303 (0.5882)
  Wk32,n=104,97,na,na,33,30,21,19,87,17,17 | -0.358 (0.4964) | -0.505 (0.5759) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -0.284 (0.4627) | -0.300 (0.5039) | -0.679 (0.5414) | -0.546 (0.5998) | -0.741 (0.6909) | -0.228 (0.5612) | -0.375 (0.7315)
  Wk36,n=102,93,na,na,30,30,21,19,84,18,16, | -0.339 (0.5687) | -0.430 (0.5573) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -0.368 (0.5397) | -0.383 (0.4500) | -0.607 (0.5538) | -0.474 (0.6032) | -0.756 (0.6844) | -0.285 (0.5891) | -0.430 (0.6723)
  Wk40,n=96,89,na,na,28,28,21,19,84,15,17 | -0.424 (0.5967) | -0.440 (0.5416) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -0.522 (0.6805) | -0.391 (0.5446) | -0.571 (0.5736) | -0.539 (0.6998) | -0.763 (0.6750) | -0.242 (0.6312) | -0.390 (0.6523)
  Wk44,n=97,90,na,na,28,27,20,18,84,15,16 | -0.331 (0.5871) | -0.449 (0.5427) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -0.277 (0.6377) | -0.523 (0.6587) | -0.638 (0.5144) | -0.514 (0.7752) | -0.781 (0.7252) | -0.308 (0.6319) | -0.203 (0.7917)
  Wk48,n-94,89,na,na,28,26,19,19,76,12,14 | -0.303 (0.5062) | -0.483 (0.5459) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -0.348 (0.5886) | -0.413 (0.5698) | -0.605 (0.6113) | -0.454 (0.5547) | -0.798 (0.6481) | -0.229 (0.6546) | -0.286 (0.7618)
  Wk52,n=92,87,na,na,28,26,20,18,79,15,15 | -0.341 (0.5428) | -0.516 (0.6036) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -0.402 (0.5436) | -0.351 (0.6335) | -0.606 (0.6492) | -0.569 (0.7126) | -0.788 (0.6853) | -0.392 (0.5216) | -0.258 (0.8298)

9. Secondary Outcome: Change From Baseline in Disease Activity Score Utilizing CRP (DAS28-CRP) - Using MMRM
Description: as for outcome 2
Time Frame: baseline, weeks 1, 2, 4, 8, 12, 16, 20 and 24
Population: Participants from the full analysis set were considered for the analysis. For Placebo and Abatacept participants, data collected after treatment switch was treated as missing, as were missing values for all treatment groups
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | AIN457 10mg/kg - 75 mg | AIN457 10mg/kg - 150 mg | Placebo | Abatacept
Number analyzed (Participants) | 138 | 137 | 138 | 39
score on a scale
  week 1, n=131,129,130,129 | -0.89 (0.069) | -0.73 (0.069) | -0.22 (0.069) | -0.50 (0.069)
  week 2, n=131,127,132,133 | -0.96 (0.080) | -0.90 (0.081) | -0.35 (0.080) | -0.78 (0.080)
  week 4, n=130,131,138,138 | -1.20 (0.090) | -1.11 (0.090) | -0.48 (0.090) | -1.11 (0.091)
  week 8, n=130,126,130,130 | -1.21 (0.093) | -1.23 (0.094) | -0.61 (0.093) | -1.55 (0.093)
  week 12, n=130,114,123,128 | -1.23 (0.097) | -1.36 (0.102) | -0.73 (0.100) | -1.78 (0.098)
  week 16, n=126,116,114,127 | -1.23 (0.108) | -1.40 (0.112) | -0.57 (0.112) | -1.71 (0.108)
  week 20, n=121,114,47,92 | -1.44 (0.108) | -1.49 (0.111) | -0.89 (0.146) | -1.96 (0.117)
  week 24, n=116,108,44,84 | -1.47 (0.115) | -1.47 (0.119) | -1.02 (0.163) | -2.07 (0.128)

10. Secondary Outcome: Change From Baseline in Disease Activity Score Utilizing CRP (DAS28-CRP) - Observed Data
Description: The DAS28 is a measure of disease activity in RA based on Swollen and Tender Joint Counts (out of a total of 28), hsCRP and the Patient's Global Assessment of Disease Activity. A DAS28 score greater than 5.1 implies active disease, equal to or less than 3.2 low disease activity, and less than 2.6 remission. A negative change from baseline indicates improvement. The DAS28-CRP results from baseline up to week 52 were based on observed data, i.e. without imputation.
Time Frame: baseline, weeks 1, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AIN457 10mg/kg - 75 mg | AIN457 10mg/kg - 150 mg | Placebo | Abatacept | Placebo Non-responder - AIN457 75mg | Placebo Non-responder - AIN457 150mg | Placebo Responder - AIN457 75mg | Placebo Responder - AIN457 150mg | Abatacept Responders | Abatacept Non-responders - AIN457 75mg | Abatacept Non-responders - AIN457 150mg
Number analyzed (Participants) | 138 | 137 | 138 | 39 | 39 | 23 | 22 | 138 | 101 | 18 | 19
score on a scale
  Wk1,n=131,129,130,129,39,35,21,22, 95,17,17 | -0.886 (0.9784) | -0.759 (0.8654) | -0.211 (0.6877) | -0.502 (0.7539) | -0.147 (0.5527) | -0.141 (0.7095) | -0.572 (0.7856) | -0.235 (0.7699) | -0.577 (0.7924) | -0.361 (0.3578) | -0.222 (0.7695)
  Wk2,n=131,127,132,133,39,36,23,21,98,17,18 | -0.909 (1.0331) | -0.900 (1.0284) | -0.363 (0.8388) | -0.755 (0.9234) | -0.191 (0.7331) | -0.368 (0.7170) | -0.835 (0.9466) | -0.292 (0.7448) | -0.755 (0.9234) | -0.882 (0.9526) | -0.359 (0.8980)
  Wk4,n=130,131,129,128,39,38,23,21,92,17,19 | -1.163 (1.1656) | -1.150 (1.1942) | -0.492 (0.8876) | -1.095 (1.0483) | -0.252 (0.8116) | -0.352 (0.7471) | -1.034 (0.9119) | -0.767 (0.9661) | -1.268 (1.0533) | -0.595 (1.1160) | -0.706 (0.6999)
  Wk8,n=130,126,130,130,39,39,23,22,94,17,19 | -1.181 (1.1821) | -1.283 (1.1678) | -0.644 (1.1356) | -1.541 (1.1172) | -0.546 (1.1597) | -0.312 (0.9151) | -1.403 (1.2060) | -0.613 (0.9772) | -1.816 (1.0708) | -0.834 (1.1469) | -0.808 (0.6444)
  Wk12,n=130,114,123,128,39,37,23,21,93,17,18 | -1.229 (1.1782) | -1.402 (1.2182) | -0.742 (1.2330) | -1.790 (1.2356) | -0.311 (0.9514) | -0.383 (1.1765) | -1.588 (0.9714) | -1.330 (1.4721) | -2.144 (1.1028) | -0.749 (1.0757) | -0.945 (1.1008)
  Wk16,n=126,116,114,128,36,36,21,21,94,15,19 | -1.225 (1.2866) | -1.455 (1.3489) | -0.592 (1.2557) | -1.691 (1.2979) | 0.128 (0.8579) | 0.045 (0.9145) | -2.008 (0.8675) | -1.503 (0.8746) | -2.159 (1.0767) | -0.490 (0.8170) | -0.322 (1.0262)
  Wk20,n=121,114,,119,125,38,37,23,21,90,16,19 | -1.427 (1.3266) | -1.569 (1.2361) | -1.164 (1.2087) | -1.840 (1.4144) | -0.683 (1.1231) | -0.937 (1.0966) | -2.108 (1.0368) | -1.399 (1.1487) | -2.317 (1.2549) | -0.402 (0.9820) | -0.792 (1.0272)
  Wk24,n=116,108,116,117,37,36,21,22,84,15,18 | -1.467 (1.3116) | -1.579 (1.3221) | -1.248 (1.2915) | -1.989 (1.4717) | -0.666 (0.9983) | -1.140 (1.1954) | -2.343 (1.2649) | -1.362 (1.2999) | -2.435 (1.3266) | -0.772 (1.1656) | -0.923 (1.2560)
  Wk28,n=115,103,na,na,33,35,21,21,86,17,18 | -1.484 (1.3216) | -1.819 (1.3434) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -1.172 (1.1602) | -1.244 (1.2433) | -2.117 (0.8573) | -1.782 (1.0655) | -2.470 (1.2153) | -1.137 (1.2050) | -0.973 (1.1034)
  Wk32,n=103,97,na,na,33,39,23,22,87,17,16 | -1.738 (1.2783) | -1.966 (1.1770) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -1.408 (1.3855) | -1.475 (1.1846) | -2.363 (1.0711) | -1.875 (0.9807) | -2.629 (1.3104) | -0.961 (1.0043) | -1.464 (1.2025)
  Wk36,n=101,92,na,na,30,30,21,20,84,18,15 | -1.737 (1.4592) | -1.820 (1.2500) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -1.271 (1.4949) | -1.444 (1.1949) | -2.269 (1.0688) | -1.784 (0.9029) | -2.642 (1.4305) | -1.200 (1.3228) | -1.425 (0.9247)
  Wk40,n=96,90,na,na,28,28,21,19,84,15,17 | -1.742 (1.3259) | -1.788 (1.1333) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -1.354 (1.3590) | -1.494 (1.3243) | -2.315 (1.0773) | -2.134 (1.0405) | -2.549 (1.3305) | -1.201 (1.5293) | -1.612 (1.1839)
  Wk44,n=96,88,na,na,28,27,20,18,84,15,16 | -1.764 (1.3227) | -1.932 (1.2850) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -1.168 (1.2638) | -1.858 (1.2373) | -2.155 (0.9488) | -2.121 (1.1347) | -2.697 (1.2117) | -0.881 (1.3337) | -1.528 (1.2973)
  Wk48,n=94,88,na,na,28,26,18,19,76,12,14 | -1.761 (1.3152) | -2.200 (1.3293) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -1.516 (1.0635) | -1.660 (1.1805) | -2.259 (1.1813) | -1.964 (1.3404) | -2.634 (1.2189) | -1.013 (1.1738) | -1.400 (1.1985)
  Wk52,n=92,86,na,na,28,26,20,18,79,15,15 | -1.839 (1.3755) | -2.109 (1.4000) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -1.487 (1.0729) | -1.690 (1.2093) | -2.070 (0.9984) | -2.334 (1.1428) | -2.676 (1.3593) | -1.390 (1.1884) | -0.982 (1.1943)

11. Secondary Outcome: Change From Baseline in hsCRP - Observed Data
Description: Blood samples were obtained to identify the presence of inflammation, to determine its severity and to monitor response to treatment. A negative change from baseline indicates improvement. The hsCRP results from baseline up to week 52 were based on observed data, i.e. without imputation.
Time Frame: baseline, weeks 1, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | AIN457 10mg/kg - 75 mg | AIN457 10mg/kg - 150 mg | Placebo | Abatacept | Placebo Non-responder - AIN457 75mg | Placebo Non-responder - AIN457 150mg | Placebo Responder - AIN457 75mg | Placebo Responder - AIN457 150mg | Abatacept Responders | Abatacept Non-responders - AIN457 75mg | Abatacept Non-responders - AIN457 150mg
Number analyzed (Participants) | 138 | 137 | 138 | 138 | 39 | 39 | 23 | 22 | 101 | 18 | 19
mg/L
  Wk1,n=134,130,131,131,39,36,21,22,97,17,17 | -10.91 (30.815) | -10.31 (27.754) | -0.69 (15.521) | -5.64 (18.550) | -0.33 (10.430) | -0.84 (24.777) | -0.40 (12.244) | -1.50 (7.541) | -6.40 (20.458) | -2.92 (12.405) | -4.07 (10.811)
  Wk2,n=133,129,133,135,39,36,23,21,100,17,18 | -10.24 (33.209) | -11.51 (32.139) | -2.21 (14.501) | -6.36 (19.416) | 0.43 (15.333) | -5.48 (17.301) | -1.70 (11.170) | -4.78 (10.515) | -7.52 (20.301) | -3.84 (13.737) | -2.30 (19.035)
  Wk4,n=131,134,129,133,39,38,23,21,97,17,19 | -9.10 (20.514) | -10.76 (33.376) | -1.53 (19.311) | -6.70 (20.732) | 2.23 (23.317) | -1.94 (21.927) | -6.47 (12.458) | -1.95 (12.090) | -7.53 (22.982) | -4.42 (14.991) | -4.50 (11.029)
  Wk8,n=134,128,130,132,39,39,23,22,96,17,19 | -10.18 (33.400) | -12.94 (30.854) | -2.94 (20.601) | -8.48 (21.134) | -4.72 (18.766) | -3.28 (25.501) | 0.13 (18.061) | -1.50 (12.839) | -10.13 (22.724) | -.54 (14.849) | -4.59 (16.603)
  Wk12,n=133,119,128,131,39,39,23,22,96,17,18 | -9.41 (31.859) | -9.66 (24.298) | -0.69 (18.908) | -9.72 (25.787) | 2.11 (18.312) | -2.89 (20.763) | -2.74 (12.899) | 2.10 (22.545) | -12.17 (25.813) | -4.18 (16.024) | -1.94 (31.483)
  Wk16,n=129,120,121,131,36,38,21,21,96,16,19 | -9.97 (33.291) | -5.78 (25.418) | -1.82 (20.849) | -8.37 (22.571) | 3.92 (23.403) | -2.13 (24.422) | -5.67 (9.583) | -4.29 (13.497) | -11.25 (23.692) | -1.41 (8.810) | 0.32 (22.024)
  Wk20,n=124,116,120,127,38,37,23,21,91,17,19 | -9.19 (32.876) | -8.05 (22.394) | -3.75 (29.301) | -9.43 (23.212) | -5.33 (20.645) | -7.77 (27.581) | 3.23 (48.634) | -1.06 (15.737) | -11.59 (24.271) | -3.94 (15.716) | -3.99 (32.871)
  Wk24,n=121,113,116,120,37,36,21,22,86,16,18 | -6.90 (22.098) | -4.92 (23.075) | -6.88 (21.014) | -8.66 (21.574) | -7.06 (20.298) | -11.46 (26.373) | -6.40 (11.562) | 0.45 (18.244) | -11.72 (22.198) | -4.94 (13.605) | 2.63 (20.875)
  Wk28,n=119,110,na,na,34,35,21,21,89,17,18 | -4.94 (23.155) | -5.87 (25.885) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -4.43 (21.777) | -11.10 (27.186) | -7.97 (18.018) | 0.09 (24.933) | -12.08 (22.791) | -4.51 (14.144) | -1.70 (22.671)
  Wk32,n=107,101,na,na,34,32,20,21,87,17,16 | -8.57 (20.826) | 7.37 (24.564) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -4.34 (23.742) | -9.08 (25.867) | -5.02 (10.300) | -5.51 (14.279) | -12.83 (23.330) | -4.26 (15.329) | -7.14 (17.446)
  Wk36,n=107,98,na,na,32,31,21,20,85,18,15 | -6.60 (25.895) | -6.36 (22.571) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -4.21 (27.424) | -2.35 (37.226) | -2.73 (21.272) | -6.78 (13.940) | -12.19 (24.535) | -4.38 (14.479) | -0.47 (27.932)
  WK40,n=101,96,na,na,29,29,22,20,86,15,17 | -8.74 (22.257) | -7.09 (24.325) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -7.07 (26.156) | 2.39 (32.966) | -4.46 (22.808) | -4.73 (13.502) | -12.63 (23.788) | -2.75 (17.297) | -7.95 (18.343)
  Wk44,n=97,92,na,na,,28,28,20,19,85,15,16 | -6.59 (20.975) | -7.25 (24.681) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -6.66 (23.396) | -8.53 (19.970) | -6.50 (19.968) | -7.27 (13.887) | -12.32 (25.470) | -1.33 (4.846) | -3.69 (24.389)
  Wk48,n=97,91,na,na,28,29,20,19,79,13,14 | -6.19 (18.912) | -7.63 (21.682) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -10.49 (25.564) | -4.76 (15.784) | -1.43 (33.122) | -6.97 (13.680) | -13.90 (25.636) | -3.50 (21.343) | -4.48 (16.918)
  Wk52,n=95,92,na,na,29,28,20,18,83,16,16 | -6.68 (26.240) | -8.14 (22.149) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -4.63 (25.795) | -4.79 (22.882) | 2.95 (9.880) | -4.88 (11.707) | -11.19 (27.768) | -6.73 (14.972) | -5.78 (18.534)

12. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) - Observed Data
Description: Blood samples were obtained to monitor disease activity and response to treatment. A negative change from baseline indicates improvement. The ESR results from baseline up to week 52 were based on observed data, i.e. without imputation.
Time Frame: baseline, weeks 1, 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | AIN457 10mg/kg - 75 mg | AIN457 10mg/kg - 150 mg | Placebo | Abatacept | Placebo Non-responder - AIN457 75mg | Placebo Non-responder - AIN457 150mg | Placebo Responder - AIN457 75mg | Placebo Responder - AIN457 150mg | Abatacept Responders | Abatacept Non-responders - AIN457 75mg | Abatacept Non-responders - AIN457 150mg
Number analyzed (Participants) | 138 | 137 | 138 | 138 | 39 | 39 | 23 | 22 | 101 | 18 | 19
mm/hr
  Wk1,n=133,130,131,131,39,36,21,22,97,17,17, | -7.5 (18.74) | -8.4 (19.20) | -5.7 (15.68) | -9.5 (16.55) | -8.4 (12.65) | -1.1 (18.88) | -5.7 (14.97) | -7.1 (13.22) | -10.2 (17.11) | -7.7 (13.90) | -7.2 (16.30)
  Wk2,n=133,130,135,134,39,36,23,22,99,17,18 | -12.2 (19.06) | -10.5 (19.05) | -5.7 (18.22) | -11.0 (19.50) | -4.0 (12.69) | -5.6 (26.44) | -9.7 (17.86) | -6.6 (14.44) | -10.2 (20.33) | -12.5 (16.71) | -13.6 (17.78)
  Wk4,n=133,135,131,133,39,39,23,21,97,17,19 | -12.7 (22.23) | -12.1 (21.88) | -6.0 (18.90) | -12.6 (18.14) | -3.7 (14.35) | -3.8 (20.50) | -9.3 (13.81) | -8.2 (23.89) | -12.3 (18.66) | -15.8 (17.49) | -11.3 (16.46)
  Wk8,n=133,129,131,132,39,39,23,22,96,17,19 | -15.4 (20.38) | -15.7 (21.62) | -6.4 (22.72) | -17.6 (20.89) | -9.4 (19.24) | -0.9 (27.25) | -8.2 (24.09) | -8.3 (14.29) | -18.3 (21.56) | -13.9 (23.29) | -17.6 (15.03)
  Wk12,n=133,118,127,131,39,39,23,21,96,17,18 | -14.7 (20.08) | -18.4 (21.18) | -5.8 (21.02) | -19.4 (20.97) | -5.9 (17.96) | -1.5 (25.62) | -11.2 (18.06) | -5.5 (20.06) | -19.9 (21.08) | -18.4 (23.07) | -17.9 (19.31)
  Wk16,n=129,121,122,130,36,38,21,22,95,16,19 | -16.2 (21.22) | -15.6 (19.09) | -6.5 (23.48) | -18.5 (24.32) | -3.1 (19.21) | -1.1 (25.47) | -17.6 (23.03) | -4.9 (20.54) | -21.1 (24.73) | -14.9 (17.78) | -8.8 (25.22)
  Wk20,n=123,116,120,127,38,37,23,21,91,17,19 | -16.3 (20.90) | -17.7 (19.90) | -9.1 (26.29) | -21.1 (23.66) | -21.1 (23.66) | -10.5 (20.08) | -7.4 (29.40) | -11.6 (34.23) | -7.0 (22.32) | -22.0 (23.60) | -20.5 (22.81)
  Wk24,n=122,113,117,123,38,36,21,22,88,17,18 | -13.9 (23.65) | -16.0 (20.20) | -12.0 (24.31) | -19.6 (24.52) | -10.8 (20.33) | -14.7 (27.77) | -16.1 (21.57) | -5.5 (27.07) | -21.1 (24.62) | -20.7 (20.65) | -11.4 (26.96)
  Wk28,n=119,110,na,na,34,35,21,21,89,17,19 | -15.4 (22.95) | -16.8 (23.05) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -17.9 (24.87) | -12.5 (30.87) | -12.3 (24.10) | -14.6 (17.31) | -22.4 (22.90) | -26.1 (19.83) | -17.4 (24.77)
  Wk32,n=108,101,na,na,34,32,21,21,88,17,16 | -18.3 (23.51) | -17.4 (21.57) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -17.2 (16.70) | -12.8 (26.21) | -16.8 (24.37) | -14.1 (20.72) | -25.5 (24.89) | -25.7 (21.14) | -23.1 (21.46)
  Wk36,n=107,98,na,na,32,31,21,20,87,18,16 | -16.6 (25.20) | -18.4 (21.51) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -17.8 (21.72) | -13.4 (29.49) | -17.3 (22.02) | -16.5 (17.95) | -21.7 (25.40) | -26.0 (21.21) | -16.6 (23.31)
  Wk40,n=101,96,na,na,29,29,22,20,85,15,17 | -18.1 (21.06) | -17.3 (21.05) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -20.6 (19.66) | -12.3 (26.37) | -13.3 (18.78) | -16.4 (21.79) | -22.2 (26.24) | -23.8 (22.96) | -22.9 (15.57)
  Wk44,n=98,93,na,na,28,28,20,19,85,15,16 | -18.0 (21.08) | -16.7 (23.87) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -20.1 (17.61) | -16.0 (25.30) | -12.0 (29.20) | -19.2 (22.57) | -24.9 (25.66) | -22.3 (23.36) | -18.5 (21.00)
  Wk48,n=97,92,na,na,28,30,20,19,79,13,14 | -17.8 (23.11) | -19.8 (20.30) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -20.8 (18.26) | -7.2 (22.58) | -12.2 (29.55) | -19.4 (20.58) | -23.9 (25.56) | -18.9 (26.41) | -20.2 (18.16)
  Wk52,n=94,91,na,na,29,28,20,18,83,16,16 | -17.7 (21.08) | -20.6 (23.48) | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | NA (NA) — After week 24, placebo and abatacept analysis was done on 'AIN457 switch' groups only. | -14.9 (20.53) | -15.1 (21.50) | -14.4 (24.54) | -13.6 (27.16) | -25.2 (27.88) | -27.4 (22.71) | -15.4 (22.53)

ADVERSE EVENTS:
Groups:
- Any AIN457 75 mg: Any AIN457 75 mg
- Any AIN457 150 mg: Any AIN457 150 mg
Arm/Group | Any AIN457 75 mg | Any AIN457 150 mg | Placebo | Abatacept
Serious Adverse Events (participants affected / at risk) | 30/218 | 28/215 | 7/139 | 9/137
Other Adverse Events (participants affected / at risk) | 144/218 | 146/215 | 51/139 | 78/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 75 mg (N=218) | Any AIN457 150 mg (N=215) | Placebo (N=139) | Abatacept (N=137)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Cyst (General disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0
Device dislocation (General disorders) | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Eye abscess (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 0 | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster oticus (Infections and infestations) | 0 | 1 | 0 | 0
Joint abscess (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural headache (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Acquired claw toe (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Formication (Nervous system disorders) | 1 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Meningorrhagia (Nervous system disorders) | 1 | 0 | 0 | 0
Perineurial cyst (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 1 | 0 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 75 mg (N=218) | Any AIN457 150 mg (N=215) | Placebo (N=139) | Abatacept (N=137)
Anaemia (Blood and lymphatic system disorders) | 10 | 10 | 8 | 6
Leukopenia (Blood and lymphatic system disorders) | 6 | 4 | 0 | 2
Lymphopenia (Blood and lymphatic system disorders) | 5 | 5 | 4 | 2
Neutrophilia (Blood and lymphatic system disorders) | 2 | 2 | 3 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 4 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 5 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 16 | 12 | 0 | 9
Dyspepsia (Gastrointestinal disorders) | 6 | 3 | 1 | 2
Nausea (Gastrointestinal disorders) | 9 | 5 | 2 | 1
Oedema peripheral (General disorders) | 9 | 6 | 0 | 2
Pyrexia (General disorders) | 3 | 9 | 1 | 2
Bronchitis (Infections and infestations) | 10 | 12 | 0 | 5
Gastroenteritis (Infections and infestations) | 8 | 4 | 0 | 5
Influenza (Infections and infestations) | 7 | 13 | 1 | 1
Nasopharyngitis (Infections and infestations) | 24 | 17 | 4 | 8
Oral candidiasis (Infections and infestations) | 1 | 3 | 0 | 4
Pharyngitis (Infections and infestations) | 10 | 5 | 1 | 5
Respiratory tract infection (Infections and infestations) | 2 | 5 | 0 | 1
Rhinitis (Infections and infestations) | 8 | 12 | 1 | 3
Sinusitis (Infections and infestations) | 9 | 7 | 2 | 1
Tonsillitis (Infections and infestations) | 6 | 3 | 0 | 0
Tracheobronchitis (Infections and infestations) | 5 | 1 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 18 | 21 | 9 | 6
Urinary tract infection (Infections and infestations) | 16 | 10 | 2 | 8
Viral infection (Infections and infestations) | 1 | 6 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 5 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 7 | 3 | 1
Alanine aminotransferase increased (Investigations) | 4 | 3 | 0 | 3
Lipoprotein (a) increased (Investigations) | 2 | 6 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 5 | 3 | 1 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 | 7 | 6 | 10
Hyperlipidaemia (Metabolism and nutrition disorders) | 6 | 11 | 2 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 | 2 | 3 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 3 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 15 | 1 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 5 | 5 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 10 | 2 | 6
Bursitis (Musculoskeletal and connective tissue disorders) | 6 | 5 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 7 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 4 | 0 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 19 | 22 | 6 | 6
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 | 5 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 0 | 3
Headache (Nervous system disorders) | 18 | 11 | 4 | 9
Paraesthesia (Nervous system disorders) | 3 | 5 | 1 | 1
Insomnia (Psychiatric disorders) | 3 | 4 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 5 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 5 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 7 | 4 | 1 | 3
Hypertension (Vascular disorders) | 20 | 10 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.